CLINICAL TRIAL: NCT04204772
Title: A Pilot Feasibility Study of Activated Charcoal in Healthy Adult Volunteers
Brief Title: A Pilot Feasibility Study of Activated Charcoal in Healthy Volunteers
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 2019LS014; HM2019-12 (Other: University of Minnesota Masonic Cancer Center); UL1TR002494 (NIH)
Record Dates: First submitted 2019-12-17; First posted 2019-12-19 (Actual); Results first posted 2023-10-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Healthy Adult Volunteers
Keywords: activated charcoal
MeSH Terms: conditions — Anthrax | interventions — Charcoal

STUDY DESIGN:
Intervention Model Description: 12 healthy volunteers will be enrolled to determine the two most palatable and tolerable AC combinations. There will be a total of 4 combinations (2 AC doses and 2 solutions) in stage 1. Each participant will drink an assigned combination every day for 3 consecutive days (Monday, Tuesday, Wednesday, "M/T/W") and switch to a different assigned combination M/T/W the following week. AC solution assignments will be defined before the study using a balanced incomplete block design
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Solution A Dose 1, Then Solution B Dose 2 (Experimental): Participants initially assigned to Solution A Dose 1 will complete the three day course (days 1-3) and switch to the Solution B Dose 2 arm to complete the three day course (days 8-10). The dose level for Solution A Dose 1 is 12 grams of medical grade oral AC mixed with 4 ounces of tap water. Participants will report on a daily basis and consume the assigned combination of oral AC.
  Interventions: Biological: Activated charcoal and Tap Water
- Solution A Dose 2, Then Solution B Dose 1 (Experimental): Participants initially assigned to Solution A Dose 2 will complete the three day course (days 1-3) and switch to the Solution B Dose 1 arm to complete the three day course (days 8-10). The dose level for Solution A Dose 2 is 25 grams of medical grade oral AC mixed with 4 ounces of tap water. Participants will report on a daily basis and consume the assigned combination of oral AC.
  Interventions: Biological: Activated charcoal and Tap Water
- Solution B Dose 1, Then Solution A Dose 2 (Experimental): Participants initially assigned to Solution B Dose 1 will complete the three day course (days 1-3) and switch to the Solution A Dose 2 arm to complete the three day course (days 8-10). The dose level for Solution B Dose 1 is 12 grams of medical grade oral AC mixed with 4 ounces of apple juice. Participants will report on a daily basis and consume the assigned combination of oral AC.
  Interventions: Biological: Activated Charcoal and Apple Juice
- Solution B Dose 2, Then Solution A Dose 1 (Experimental): Participants initially assigned to Solution B Dose 2 will complete the three day course (days 1-3) and switch to the Solution A Dose 1 arm to complete the three day course (days 8-10). The dose level for Solution B Dose 2 is 25 grams of medical grade oral AC mixed with 4 ounces of apple juice. Participants will report on a daily basis and consume the assigned combination of oral AC.
  Interventions: Biological: Activated Charcoal and Apple Juice

INTERVENTIONS:
Biological: Activated charcoal and Tap Water — 12 grams of AC mixed with Tap water or 25 grams of AC mixed with Tap water
  Other Names: Medical grade AC, "Activated Charcoal Powder, USP", activated carbon.
  Arms: Solution A Dose 1, Then Solution B Dose 2; Solution A Dose 2, Then Solution B Dose 1
Biological: Activated Charcoal and Apple Juice — 12 grams of AC with Apple Juice or 25 grams of AC with Apple Juice
  Arms: Solution B Dose 1, Then Solution A Dose 2; Solution B Dose 2, Then Solution A Dose 1

SUMMARY:
This is a pilot study designed to test feasibility, tolerability, and safety of medical grade oral Activated Charcoal (AC) in 12 healthy volunteers. To determine the two most palatable and tolerable AC combinations. There will be a total of 4 combinations (2 AC doses and 2 solutions) in stage 1. Each participant will drink an assigned combination every day for 3 consecutive days (Monday, Tuesday, Wednesday, "M/T/W") and switch to a different assigned combination M/T/W the following week. AC solution assignments will be defined before the study using a balanced incomplete block design. Each subject will rate their experience using a 5-point scale every day for the 12 days they are on study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* No use of prescription medications, including oral birth control, currently or in the last 30 days
* Sexually active women must be using an effective form of contraception. Note that subjects who are on oral contraception should use an additional form of contraception such as barrier methods, as AC may interfere with the efficacy of oral contraceptive
* Voluntary written consent signed before performance of any study-related procedure

Exclusion Criteria:

* At risk of GI hemorrhage or perforation due to underlying pathology, recent surgery, or medical conditions that could be adversely affected by the administration of AC
* Planning to have an endoscopic procedure
* Known hypersensitivity to AC
* Non-English speakers

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-01-22 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Armin Rashidi, MD, PhD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy Volunteers will respond to poster advertisements containing a brief study description and the contact information of the study coordinator.
Pre-assignment Details: Participants were given dose assignments at the time of study registration using a balanced incomplete block design. One participant was assigned two out of the four possible solution-doses. Each participant will drink an assigned combination every day for 3 consecutive days (Monday, Tuesday, Wednesday, "M/T/W") and switch to a different assigned combination M/T/W the following week.
Period: Overall Study
Arm/Group | Solution A Dose 1, Then Solution B Dose 2 | Solution A Dose 2, Then Solution B Dose 1 | Solution B Dose 1, Then Solution A Dose 2 | Solution B Dose 2, Then Solution A Dose 1
Started | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Solution A Dose 1, Then Solution B Dose 2 | Solution A Dose 2, Then Solution B Dose 1 | Solution B Dose 1, Then Solution A Dose 2 | Solution B Dose 2, Then Solution A Dose 1 | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 3 | 3 | 12
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 1 | 0 | 4
  Male | 1 | 2 | 2 | 3 | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 3 | 3 | 12

OUTCOME MEASURES:

1. Primary Outcome: Average Palatability Rating
Description: Each healthy volunteer will rate their experience using a 5-point scale (1=terrible, 2=bad, 3=okay, 4=good, 5=great) every day.
Time Frame: two weeks
Measure: Mean (Standard Deviation); unit: score on a scale out of 5
Groups:
- Solution A Dose 1: The dose level for Solution A Dose 1 is 12 grams of medical grade oral AC mixed with 4 ounces of tap water. Participants will report on a daily basis and consume the assigned combination of oral AC.
- Solution A Dose 2: The dose level for Solution A Dose 2 is 25 grams of medical grade oral AC mixed with 4 ounces of tap water. Participants will report on a daily basis and consume the assigned combination of oral AC.
- Solution B Dose 1: The dose level for Solution B Dose 1 is 12 grams of medical grade oral AC mixed with 4 ounces of apple juice. Participants will report on a daily basis and consume the assigned combination of oral AC.
- Solution B Dose 2: The dose level for Solution B Dose 2 is 25 grams of medical grade oral AC mixed with 4 ounces of apple juice. Participants will report on a daily basis and consume the assigned combination of oral AC.
Arm/Group | Solution A Dose 1 | Solution A Dose 2 | Solution B Dose 1 | Solution B Dose 2
Number analyzed (Participants) | 6 | 6 | 6 | 6
score on a scale out of 5 | 3.5 (0.9) | 4.0 (0.8) | 4.9 (0.2) | 4.4 (0.6)

2. Secondary Outcome: Number of Participants With Grade 2 and Above Adverse Events Related to Activated Charcoal by Day 12
Time Frame: 12 days
Population: Adverse events analyzed on a per intervention basis.
Measure: Count of Participants; unit: Participants
Groups:
- Solution A Dose 1: Participants initially assigned to Solution A Dose 1 will complete the three day course and switch to the second assigned Solution arm to complete the second three day course . The dose level for Solution A Dose 1 is 12 grams of medical grade oral AC mixed with 4 ounces of tap water. Participants will report on a daily basis and consume the assigned combination of oral AC. Participant adverse events recorded on a per intervention basis.
- Solution A Dose 2: Participants initially assigned to Solution A Dose 2 will complete the three day course and switch to the second assigned Solution arm to complete the second three day course. The dose level for Solution A Dose 2 is 25 grams of medical grade oral AC mixed with 4 ounces of tap water. Participants will report on a daily basis and consume the assigned combination of oral AC. Participant adverse events recorded on a per intervention basis.
- Solution B Dose 1: Participants initially assigned to Solution B Dose 1 will complete the three day course and switch to the second assigned Solution arm to complete the second three day course. The dose level for Solution B Dose 1 is 12 grams of medical grade oral AC mixed with 4 ounces of apple juice. Participants will report on a daily basis and consume the assigned combination of oral AC. Participant adverse events recorded on a per intervention basis.
- Solution B Dose 2: Participants initially assigned to Solution B Dose 2 will complete the three day course and switch to the second assigned Solution arm to complete the second three day course. The dose level for Solution B Dose 2 is 25 grams of medical grade oral AC mixed with 4 ounces of apple juice. Participants will report on a daily basis and consume the assigned combination of oral AC. Participant adverse events recorded on a per intervention basis.
Arm/Group | Solution A Dose 1 | Solution A Dose 2 | Solution B Dose 1 | Solution B Dose 2
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Participants were contacted during the first two weeks for any AEs.
Description: Adverse events collected on a whole trial basis.
Groups:
- Solution A Dose 1: Participants initially assigned to Solution A Dose 1 will complete the three day course (days 1-3) and switch to the Solution B Dose 2 arm to complete the three day course (days 8-10). The dose level for Solution A Dose 1 is 12 grams of medical grade oral AC mixed with 4 ounces of tap water. Participants will report on a daily basis and consume the assigned combination of oral AC.
- Solution A Dose 2: Participants initially assigned to Solution A Dose 2 will complete the three day course (days 1-3) and switch to the Solution B Dose 1 arm to complete the three day course (days 8-10). The dose level for Solution A Dose 2 is 25 grams of medical grade oral AC mixed with 4 ounces of tap water. Participants will report on a daily basis and consume the assigned combination of oral AC.
- Solution B Dose 1: Participants initially assigned to Solution B Dose 1 will complete the three day course (days 1-3) and switch to the Solution A Dose 2 arm to complete the three day course (days 8-10). The dose level for Solution B Dose 1 is 12 grams of medical grade oral AC mixed with 4 ounces of apple juice. Participants will report on a daily basis and consume the assigned combination of oral AC.
- Solution B Dose 2: Participants initially assigned to Solution B Dose 2 will complete the three day course (days 1-3) and switch to the Solution A Dose 1 arm to complete the three day course (days 8-10). The dose level for Solution B Dose 2 is 25 grams of medical grade oral AC mixed with 4 ounces of apple juice. Participants will report on a daily basis and consume the assigned combination of oral AC.
Arm/Group | Solution A Dose 1 | Solution A Dose 2 | Solution B Dose 1 | Solution B Dose 2
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 3/6 | 2/6 | 3/6 | 3/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Solution A Dose 1 (N=6) | Solution A Dose 2 (N=6) | Solution B Dose 1 (N=6) | Solution B Dose 2 (N=6)
abdominal fullness/bloating (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) — AEs were all grade 1 and included abdominal fullness/bloating in 4 (33%) subjects, abdominal pain in 4 (33%) subjects, nausea in 2 (17%) subjects, constipation in 2 (17%) subjects, and diarrhea in 1 (8%) subject.
abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) — AEs were all grade 1 and included abdominal fullness/bloating in 4 (33%) subjects, abdominal pain in 4 (33%) subjects, nausea in 2 (17%) subjects, constipation in 2 (17%) subjects, and diarrhea in 1 (8%) subject.
nausea (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) — AEs were all grade 1 and included abdominal fullness/bloating in 4 (33%) subjects, abdominal pain in 4 (33%) subjects, nausea in 2 (17%) subjects, constipation in 2 (17%) subjects, and diarrhea in 1 (8%) subject.
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) — AEs were all grade 1 and included abdominal fullness/bloating in 4 (33%) subjects, abdominal pain in 4 (33%) subjects, nausea in 2 (17%) subjects, constipation in 2 (17%) subjects, and diarrhea in 1 (8%) subject.
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — AEs were all grade 1 and included abdominal fullness/bloating in 4 (33%) subjects, abdominal pain in 4 (33%) subjects, nausea in 2 (17%) subjects, constipation in 2 (17%) subjects, and diarrhea in 1 (8%) subject.
Mild Throat Pain/dryness (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-10-18): https://cdn.clinicaltrials.gov/large-docs/72/NCT04204772/Prot_SAP_000.pdf
  • Informed Consent Form (2020-01-21): https://cdn.clinicaltrials.gov/large-docs/72/NCT04204772/ICF_001.pdf